CLINICAL TRIAL: NCT05749822
Title: Fenofibrate Combined With Ursodeoxycholic Acid in Compensated Cirrhosis Patients With Primary Biliary Cholangitis Who Had an Inadequate Response to Ursodeoxycholic Acid
Brief Title: Fenofibrate for Compensated Cirrhosis Patients With Primary Biliary Cholangitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20222293-C-1
Record Dates: First submitted 2022-12-29; First posted 2023-03-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-UDCA (Placebo Comparator): 1 tablet/ day and UDCA 13-15mg/kg/day for 12 months
  Interventions: Drug: Placebo; Drug: UDCA
- Fenofibrate-UDCA (Experimental): Fenofibrate 200 mg/day and UDCA 13-15mg/kg/day for 12 months
  Interventions: Drug: Fenofibrate 200mg; Drug: UDCA

INTERVENTIONS:
Drug: Fenofibrate 200mg — Fenofibrate 200mg/day
  Arms: Fenofibrate-UDCA
Drug: Placebo — 1 tablet/ day
  Arms: Placebo-UDCA
Drug: UDCA — UDCA 13-15mg/kg/day

SUMMARY:
The main objectives of the study were to assess the effects of fenofibrate on serum alkaline phosphatase, as a composite endpoint and on safety in participants with primary biliary cholangitis (PBC).

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, parallel-group study that aims to assess the efficacy and safety of fenofibrate in patients with compensated cirrhosis PBC who had an inadequate biochemical response to UDCA. Fenofibrate or placebo 200 mg will be daily administered in combination with UDCA 13-15 mg/kg/d for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have provided written informed consent
* Age 18-75 years;
* BMI 17-28 kg/m2
* Male or female with a diagnosis of PBC, by at least two of the following criteria:

  1. History of AP above ULN for at least six months;
  2. Positive AMA titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies;
  3. Documented liver biopsy result consistent with PBC.
* Diagnosis of compensated cirrhosis, as demonstrated by the presence of ≥ 1 of the following 4 diagnostic factor

  1. The histology was consistent with the diagnosis of liver cirrhosi;
  2. Endoscopy shows esophageal and gastric varices or ectopic varices of digestive tract, excluding non cirrhotic portal hypertension;
  3. Ultrasound or CT and other imaging examinations indicate the characteristics of liver cirrhosis or portal hypertension, such as splenomegaly, portal vein ≥ 1.3 cm, or liver stiffness measured by transient elastography>16.9 kPa;
  4. Abnormal laboratory inspection indicators (2 out of 4): 1) PLT < 100 × 109/L, and no other reason can be explained; 2) Serum albumin<35 g/L, excluding malnutrition or kidney disease and other causes; 3) INR > 1.3 or PT prolongation (stop thrombolytic or anticoagulant drugs for more than 7 days); 4) AST/PLT (APRI)>2）
* Incomplete response to UDCA defined by ALP > 1.67 x ULN
* Taking UDCA for at least 6 months (stable dose for ≥ 3 months) prior to Day 0

Exclusion Criteria:

* History or presence of other concomitant liver diseases.
* ALT or AST > 5×ULN, TBIL > 3×ULN.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Allergic to fenofibrate or ursodeoxycholic acid.
* Taking hepatotoxic drugs (e.g., dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than 2 weeks within 6 months, and long-term hormonal users.
* Recurrent variceal bleeding, poorly controlled hepatic encephalopathy or refractory ascites.
* Patients with a history of severe cardiac, cerebrovascular, renal, respiratory disease or functional failure, and psychiatric disorders (including those due to alcohol and drug abuse).
* Creatinine >1.5×ULN and creatinine clearance <60 ml/min.
* Currently using statins (such as pravastatin, fluvastatin, and simvastatin), other fibrates (such as gemfibrozil and bezafibrate), and drugs structurally similar to fenofibrate (like ketoprofen).
* Planned to receive an organ transplant or an organ transplant recipient.
* Needing Liver transplantation within 1 year according to the Mayo Rick score.
* Any other condition(s) that would compromise the safety of the subject or compromise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with biochemical response | 48 weeks
  The normalisation of Alkaline Phosphatase

SECONDARY OUTCOMES:
Percentage of patients having biochemical response | 4, 12, 24 and 36weeks
  The normalisation of Alkaline Phosphatase at 4, 12, 24, and 36 weeks.
Assessment of the pruritus and fatigue | 4, 12, 24, 36, and 48 weeks
  Change From Baseline in Fatigue and Pruritus as Assessed by Visual Analogue Scale (VAS) Total Score for Fatigue and Pruritus. (0-10, higher scires mean a worse outcome)
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of creatinine
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase Blood urea nitrogen
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of creatine kinase
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase ALT and AST.
Survival without transplantation and hepatic impairment | 48 weeks
  Occurrence of ascites, variceal bleeding, hepatic encephalopathy, liver-transplantation, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, Principal Investigator — Xijing Hospital, Air Force Military Medical Universit
Locations (12):
- China (12):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Xijing Hospital, Xi'an, Shaanxi
  - Yan'an University Affiliated Hospital, Yan’an, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Tianjin Medical University General Hospital, Tianjin